CLINICAL TRIAL: NCT01602627
Title: A Phase I Dose Escalation, Single Center, Open-Label Study of AUY922 Administered IV on a Once-Weekly Schedule in Adult Patients 75 Years of Age or Older With Advanced Solid Malignancies
Brief Title: Hsp90 Inhibitor AUY922 in Treating Older Patients With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dale Shepard, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Dale Shepard, MD, PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3Y10; NCI-2011-03107 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-05-16; First posted 2012-05-21 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive Hsp90 inhibitor AUY922 IV over 1 hour on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Hsp90 inhibitor AUY922; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Hsp90 inhibitor AUY922 — Given IV
  Other Names: AUY922
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of Hsp90 inhibitor AUY922 in treating older patients with advanced solid malignancies. Hsp90 inhibitor AUY922 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective is to determine the maximally tolerated dose (MTD) of AUY922 (Hsp90 inhibitor AUY922) as a single agent when administered intravenously (IV) on a once-weekly schedule to adult patients 75 years of age or older with advanced solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists.

SECONDARY OBJECTIVES:

I. To characterize the safety and tolerability of treatment with AUY922. II. To characterize the pharmacokinetic profiles of AUY922, including the parent drug and any potential metabolites.

III. To determine the efficacy of AUY922 in elderly patients with measurable disease.

IV. To evaluate of effect of geriatric-focused assessment of comorbidity and functional status on the toxicity and response to AUY922.

V. To assess the ethical constraints to enrollment of elderly patients in phase I trials.

TERTIARY OBJECTIVES:

I. Determine the effect of therapy with AUY922 on the number of circulating tumor cells (CTC).

II. To assess changes HSP70 induction as a measure of pharmacodynamic effect in pre- and post-AUY922 samples in peripheral blood mononuclear cell (PBMCs) to explore age-related differences in HSP90 inhibition by AUY922 compared with the previous phase I trial.

III. To assess changes in cellular response markers of apoptosis in pre- and post-AUY922 dosing in peripheral blood including measurement of M30 and M65 to explore age-related differences in pharmacodynamics compared to patients enrolled in the previous phase I trial.

IV. To determine associations between pharmacokinetic (PK) and pharmacodynamic (PD) parameters.

V. To determine the relationship between geriatric-focused assessment of comorbidity and functional ability and toxicity and response.

OUTLINE: This is a dose-escalation study.

Patients receive Hsp90 inhibitor AUY922 IV over 1 hour on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically proven solid tumor malignancy which is refractory to standard therapy and for which no curative therapy is available
* Patients must have at least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST); irradiated lesions are only evaluable for disease progression
* Eastern Cooperative Oncology Group (ECOG) Performance Status of =< 1
* Life expectancy of >= 12 weeks
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dl
* Platelets (plt) >= 100 x 10^9/L
* Potassium within normal limits or correctable with supplements
* Total calcium (corrected for serum albumin) and phosphorus within normal limits
* Magnesium above lower limit of normal (LLN) or correctable with supplements
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) =< 2.5 x upper limit of normal (ULN) if no liver metastases are present
* AST/SGOT and ALT/SGPT =< 5 x ULN if liver metastases are present
* Serum bilirubin =< 1.5 x ULN
* Serum creatinine =< 1.5 x ULN or 24-hour clearance >= 50 ml/min
* Patients must be able to understand and voluntarily sign written informed consent

Male participants with partners who are of child bearing potential must:

* Agree to use double barrier method of birth control 28 days prior to study entry, during course of study and for 28 days following the last dose of AUY922
* OR have history of a vasectomy

Exclusion Criteria:

Patients with central nervous system (CNS) metastasis which are:

* Symptomatic or
* Require treatment for symptom control and/or
* Growing Note: Patients without clinical signs or symptoms of CNS involvement are not required to have a computed tomography (CT)/magnetic resonance imaging (MRI) of the brain
* Prior treatment with any heat shock protein (HSP)90 or histone deacetylase (HDAC) inhibitor compounds

Patients who received systemic anti-cancer treatment prior to the first dose of AUY922 within the following time frames:

* Radiotherapy or conventional chemotherapy: within 4 weeks
* Palliative radiotherapy: within 2 weeks
* Nitrosoureas, mitomycin, or monoclonal antibodies, such as trastuzumab, within 6 weeks
* Any systemic anti-cancer treatment for which the elimination period is not known, or investigational drugs (i.e. targeted agents) within a duration of =< 5 half lives of the agent and their active metabolites (if any)
* Treatment with therapeutic doses of coumadin-type anticoagulants (maximum daily dose of 2 mg, for line patency permitted)
* Unresolved diarrhea >= Common Terminology Criteria for Adverse Events (CTCAE) grade 1, despite treatment with antidiarrheal agents
* Patients with malignant ascites that require invasive treatment
* Male patients whose partners are women of child-bearing potential (WCBP) not using double-barrier methods of contraception
* Acute or chronic liver or renal disease
* Other concurrent severe and/or uncontrolled medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol
* Major surgery =< 2 weeks prior to Cycle 1, Day 1 or who have not recovered from such therapy; (placement of a venous access device within 2 weeks is permitted)

Impaired cardiac function, including any one of the following:

* History (or family history) of long QT syndrome
* Mean corrected QT interval (QTc) >= 450 msec on baseline electrocardiogram (ECG)
* History of clinically manifested ischemic heart disease =< 6 months prior to study start
* History of heart failure or left ventricular (LV) dysfunction (left ventricular ejection fraction [LVEF] =< 45%) by multigated acquisition scan (MUGA) or echocardiogram (ECHO)
* Clinically significant ECG abnormalities including 1 or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB); ST segment elevation or depression > 1mm, or 2nd (Mobitz II), or 3rd degree atrioventricular (AV) block
* History or presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes
* Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Clinically significant resting bradycardia (< 50 beats per minute)
* Patients who are currently receiving treatment with any medication which has a relative risk of prolonging the corrected QT using Bazett's formula (QTcB) interval or inducing Torsades de Pointes and cannot be switched or discontinued to an alternative drug prior to commencing AUY922
* Patients who are dependent on a pacemaker due to cardiac conduction dysfunction; known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Patients unwilling or unable to comply with the protocol

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
MTD of Hsp90 inhibitor AUY922 | at 28 days
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as clinically relevant, and occurs < 28 days following the first dose of AUY922. Toxicity will be measured by CTCAE criteria (Version 4.02). The MTD will be determined using a standard design.

SECONDARY OUTCOMES:
Toxicity by CTCAE (v 4.02) | at 28 days
Pharmacokinetic parameters, including area under the curve (AUC), clearance, volume of distribution (VD), time to the maximum concentration (Tmax), maximum plasma concentration (Cmax), and elimination half-life | at baseline and at 28 days (first cycle)
  Prior to 1st infusion; 30 minutes after start infusion; end infusion; 5, 30 minutes post-infusion; 1, 2, 4, 5, 24, 48 hours post-infusion course 1 days 8 (pretreatment) and 15 (pretreatment/end infusion); and course 2 day 1 (pretreatment/end infusion)
Tumor response will be measured by RECIST criteria (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD], overall response [OR], response rate [RR]) | at baseline and at end of cycle 2 (8 weeks)
  Imaging with CT or MRI will be obtained at baseline (within 21 days of study Day 1) and every other cycle commencing at the end of cycle 2 (beginning of cycle 3). These scans should be schedule within 7 days of the start of the cycle. Imaging will be obtained at the end of the study.
Geriatric assessment will be made including Mini Mental Exam, Get up and Go, assessment of comorbidity, and Geriatric Depression Scale | at baseline and at end of cycle 2 (8 weeks)
  This trial will incorporate geriatric assessment to determine the relationship between functional ability or comorbidity and treatment response or toxicity. Patients will be have a geriatric assessment which will included a range of assessments, such as mini mental status, up and go test, and the geriatric depression scale, at baseline and after every 2 cycles of therapy.
Evaluation of responses to a bioethics questionnaire will be used to assess patient factors influencing enrollment in this elderly-specific phase I trial | Baseline
Number of Circulating Tumor Cells (CTC) at baseline and after treatment with Hsp90 inhibitor AUY922 | at baseline and end of treatment
  Blood will be collected for measurement of CTCs on Cycle 1 Day 1 pre-infusion, Cycle 2 Day 1 pre-infusion, Cycle 3 Day 1, pre-infusion, then Day 1 of every other cycle until the end of the study.
Level of HSP70 at baseline and after treatment with Hsp90 inhibitor AUY922 | at baseline and at 28 days (first cycle)
Level of M30 and M65 at baseline and following therapy with Hsp90 inhibitor AUY922 | at baseline and at 28 days (first cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Shepard, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States